CLINICAL TRIAL: NCT01219439
Title: Laboratory Evaluation of IVF Discarded Pathological Specimens and Media for Optimization of Techniques for Assisted Reproduction
Brief Title: Evaluation of Discarded Laboratory Pathological Specimens and Media
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-14
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Non-viable Oocytes; Extra Spermatozoa; Seminal Fluid; Granulosa Cells; Serum; Follicular Fluid; Conditioned IVF Media
Keywords: discarded pathological specimens; discarded media; IVF

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA: Non-viable oocytes, spermatozoa, granulosa cells and follicular fluid Samples without DNA: seminal fluid, serum and conditioned IVF media
Oversight: Data Monitoring Committee: No

SUMMARY:
The researchers propose to investigate the causes, incidence, and time-related events of chromosomal and physiologic abnormalities as they relate to patient diagnosis, fertility drugs utilized, and in vitro laboratory culture conditions.

DETAILED DESCRIPTION:
We propose to identify a group of parameters that have significant predictive value for assisted reproductive technology outcomes. We seek to test, standardize and implement better methods for the freezing of oocytes and sperm prior to these techniques being used in the clinical setting. We seek to develop new methods to optimize the determination of genes and chromosomes in gametes. We hope to develop new cell surgery or micromanipulation techniques (e.g. use of cell drills and lasers in order to enhance the efficiency of procedures such as ICSI, assisted hatching, biopsy) as well as other manipulations. We will test the safety and efficiency of micro fluidics and automation in the Embryology lab. This has the potential to reduce cost, human errors, temperature and physical changes. We hope to develop new methods and media and media supplements normally found in the reproductive tract that allow for higher survival of gametes in vitro. We will also test the proficiency of laboratory staff members on techniques and/or procedures performed in the in-vitro fertilization laboratory. We will perform Quality Control to review how changes in temperature and setting can effect specimens

ELIGIBILITY:
Inclusion Criteria:

none

Exclusion Criteria:

none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing infertility treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2007-07; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Methods for the freezing of ooyctes and sperm | duration of study
  To test, standardize and implement better methods for the freezing of ooyctes and sperm prior to these techniques being used in the clinical setting.

SECONDARY OUTCOMES:
New methods of gene and chromosome analysis | duration of study
  The development of new methods to optimize the determination of genes and chromosomes in gametes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Basking Ridge, New Jersey, United States